CLINICAL TRIAL: NCT05678101
Title: Transcutaneous Electrical Nerve Stimulation (TENS) Integrated Into Pants for Relief of Postoperative Pain in Orthopedic Patients
Brief Title: TENS for Relief of Postoperative Pain in Orthopedic Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Paul Ackermann, Professor, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-ORTHTENS
Record Dates: First submitted 2023-01-03; First posted 2023-01-10 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Orthopedic Disorder; Post Operative Pain; Hip Fractures; Arthroplasty, Replacement, Hip; Internal Fixation
Keywords: transcutaneous electrical nerve stimulation; Patient Global Impression of Change; numeric pain rating scale; TENS; PGIC; NRS; Post Operative Pain; Hip Fractures
MeSH Terms: conditions — Musculoskeletal Diseases; Pain, Postoperative; Hip Fractures | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This study will be a prospective, randomized, single-blinded, placebo-controlled repeated measures design.
Who Masked: Participant
Masking Description: Fifteen of the patients will be randomized to the intervention and 15 will receive placebo (non-active TENS treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TENS (Active Comparator): The Chattanooga Physio TENS (DJO Global, Vista, CA) will be applied with mixed burst / TENS alternated, which is a 30-minute long program where the stimulation frequencies of alternate in 3 second intervals, producing a combined stimulation of 80 Hz and 2 Hz. Two programs/sessions ('a' and 'b') will be applied in succession for a total of 60-minutes (one round). In total, each day will have 3 rounds.
  The energy intensity level will firstly be adjusted for 80 Hz (TENS) until a tingling sensation is felt but no discomfort, and then the procedure will be repeat for 2 Hz.
  The patient will use a pair of pants with integrated stimulation electrodes, to which the CE-marked TENS device (Chattanooga Physio, DJO Nordic, Malmö, Sweden) will be connected and used to provide pain relief, in addition to usual postoperative care.
  The TENS device will be connected to the textile electrodes of the pants which are located 5cm in front and behind the hip incision dressing respectively.
  Interventions: Device: transcutaneous electrical nerve stimulation (TENS)
- Control (Sham Comparator): The control group will also receive the TENS-pants described above with integrated stimulation electrodes, connected to TENS treatment. However, the TENS treatment to the control group will be set such that no electricity will be applied to the patient. In all other regards, the control group will follow the same protocol as the intervention group.
  Interventions: Device: Sham transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Device: transcutaneous electrical nerve stimulation (TENS) — Chattanooga Physio TENS (DJO Global, Vista, CA)
  Other Names: electrical nerve stimulation
  Arms: TENS
Device: Sham transcutaneous electrical nerve stimulation (TENS) — Sham treatment with Chattanooga Physio TENS (DJO Global, Vista, CA)
  Arms: Control

SUMMARY:
To ensure early mobilization, minimize suffering, and to prevent postoperative complications postoperative pain should be reduced as soon and as effectively as possible.

A non-pharmacological post-operative intervention in terms of the application of transcutaneous electrical nerve stimulation (TENS), could have the potential to accelerate early mobilization and reduce the use of opioids.

The overall aim is to demonstrate that the addition of TENS to standard postoperative pain management of orthopedic patients can alleviate pain during mobilization and at rest as well as reduce opioid consumption.

DETAILED DESCRIPTION:
Hip fracture is most often addressed surgically (Allahabadi et al., 2022; RikshÖFt, 2020), and is commonly associated with a short-term increase in mortality, and long-term reduction in health-related quality of life (Alexiou et al., 2018; Dyer et al., 2016; Gjertsen et al., 2016; Griffin et al., 2015). A large part of this reduction in quality of life can be related to pain and mobility. According to the Swedish National Hip Fracture Registry (RikshÖFt, 2020), 5.8% of the patients registered in 2019 were experiencing severe pain either constantly or during activity at the 4-month follow-up; 42% were experiencing tolerable pain during activity, and 35% were pain-free.

In the larger context of Chronic PostOperative Pain (CPOP), severe pain on postoperative day 1 constitutes an important risk factor (Fletcher et al., 2015). A 10% increase in the amount of time spent in severe pain on postoperative day 1 has been associated with a 30% increase in the incidence of CPOP at a 12-month follow-up. Yet, a 2021 review on the prevention of CPOP (Carley et al., 2021) reported that there were no pharmaceutical pain treatments that could be universally or specifically recommended to reduce the incidence of CPOP.

To effectively manage acute and chronic pain disorders, Transcutaneous Electrical Nerve Stimulation (TENS) has been viewed a safe nonpharmacological addition to standard care (Jafra et al., 2022; Johnson et al., 2022; Vance et al., 2022). Conventional TENS with high frequency (50-100Hz) activates non-noxious afferents considered to inhibit nociceptive transmission at the spinal cord level, i.e., peripheral gate-control. Mixed-frequency TENS adds a low-frequency (mostly 2-10Hz) stimulation that activates small-diameter, high-threshold peripheral afferents considered to trigger brainstem opioid descending pain inhibitory pathways, i.e., central gate-control. Studies have indicated mixed-frequency TENS may be effective to mitigate post-operative pain (Bjordal, Johnson, & Ljunggreen, 2003; Hamza et al., 1999).

A non-pharmacological post-operative intervention in terms of the application of transcutaneous electrical nerve stimulation (TENS), could have the potential to accelerate early mobilization and reduce the use of opioids.

A 2019 study (Elboim-Gabyzon, Najjar, & Shtarker, 2019) demonstrated pain reduction during activity - but not at rest - following hip fracture with a 30-minute TENS intervention daily on the first 5 postoperative days. A more recent (and currently unpublished) study using TENS integrated in TENS-pants (Opolka et al., 2024) demonstrated pain reduction at rest and during activity with a single 2.5-hour intervention carried out around postoperative day 1 (POD1). However, there is there is still a lack of knowledge regarding the possible effect of a longer TENS intervention repeated over several days. Moreover, there is still a lack of statistical evidence for the opioid sparing effect of TENS following hip fracture surgery.

The primary aim of this study is to assess pain reduction and patient global impression of change following mixed-frequency TENS treatment (or placebo TENS) at rest and during activity on postoperative days 1 to 3, following hip fracture surgery. A secondary aim is to assess improvement in mobility and to test the opioid-sparing effect associated with TENS treatment. Moreover, to simplify TENS application, empower the elderly patients and improve compliance during mobilization, the authors chose to administer TENS using wearable TENS-pants with modular textile electrodes. We hypothesize that a mixed-frequency TENS intervention, carried out on POD1 to POD3, with a daily treatment duration of 3 hours, can lead to a significant opioid sparing effect, more durable pain reduction, and improve the patients' overall perception and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and above.
* Patient has undergone hip fracture surgery.
* Must be cognitively adequate.
* Must be without terminal illness.

Exclusion Criteria:

* Pregnancy
* Skin wounds
* Pacemaker
* Intracardiac defibrillator
* Ongoing thrombolysis or thromboprophylaxis.
* Class 3 and 4 heart disease
* Difficulties to understand the Swedish language
* Drug and narcotic abuses
* Postoperative delirium syndrome
* Epidural catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain estimation during rest | During intervention. Mesaured twice per round: First before mobility testing and TENS-session 'a' and a second time during the last 5 minutes of the TENS-session 'a' during inactivity.
  A 11-point numeric pain rating scale (Minimum 0, Maximum 10, higher score means worse outcome, i.e more pain) assessment will be performed during inactivity
Patient Global Impression of Change (PGIC) | During intervention. Measured twice per round after both TENS-session 'a' and 'b' respectively.
  The patient's belief about the efficacy of treatment, which ranged from 1 (minimum, "no change") to 7 (maximum, "a great deal better") will be assessed by PGIC.
Pain estimation during activity | During intervention. Measured twice per round: First after mobility testing and before TENS-session 'a' and a second time in the last 5 minutes of TENS-session 'b'.
  A 11-point numeric pain rating scale (Minimum 0, Maximum 10, higher score means worse outcome, i.e more pain) assessment will be performed during activity after the Standardized three-meter Walking test (WALK3m)

SECONDARY OUTCOMES:
Mobility testing (Walking test) | During intervention. Performed and measured twice per round: once before TENS-session 'a' and a second time during the last 5 minutes of TENS-session 'b'.
  The Standardized three-meter Walking test (WALK3m). With a stopwatch, the patient will be instructed to walk a 3 meters distance beginning from a marked position, in comfortable steps, to a stop position, turn around and walk back to the marked position where he or she started. The timing will begin when the patient starts on the word go, and the timing will end when the patient stopped at the marked position where they started. Patients will be asked whether or not they were mobilized prior to the intervention.
Analgesic consumption | During intervention. The information will be logged at the end of each day of intervention.
  Extra analgesic consumption will be documented to assess and evaluate the effect of the intervention during the following: (1) Only intervention (POD 1,2, and 3). In each day there will be three 30x2-minute long rounds of TENS-application with two interposed 30-minute breaks equalling 4 hours x 3 = 12 hours. (2) Totally during post-operative days 1, 2, and 3 equalling 24 x 3 = 72 hours.
Mobility testing (Put on pants time) | During intervention. Measured once per day: Before the first pain assessment during rest and before TENS-session 'a' of the first round.
  At the start of each day, before the first intervention round the duration of putting on the TENS-pants will be logged. The timer will start once the first NRS at rest has been taken and the TENS-pants are ready to be applied to the patient and it will stop once the pants are worn and ready for TENS-application.
Patients-reported impression of TENS (Qualitative assessment) | Immediately after intervention
  A short follow-up will be performed after the intervention.
  The patients in both active and placebo groups will be asked to answer a questionnaire on their attitude toward TENS and the intervention. Answers will be provided on a five-level Likert-type scale on the following statements:
  1. I think TENS therapy is comfortable for me.
  2. I would like to use TENS again if I were to undergo another surgery in the future.
  3. I think the TENS-pants were comfortable to wear.
  4. I would feel confident to put on and take off the TENS-pants by myself.
  5. I would feel confident to put on and take off the TENS-pants with the help of a family member or care assistant.
  6. If you ever need to use TENS-PANTS at home, would you prefer to use "diaper-like" pants or "normal" pants?
  In addition, patients will be asked to provide free-form general comments on the product and study.

CONTACTS AND LOCATIONS:
Overall Officials: Paul W Ackermann, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska university Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared on personal application with good reasoning.
Supporting Information: Study Protocol, SAP
Time Frame: During 2025.
Access Criteria: On reasonable request

REFERENCES:
- [Derived] Opolka Y, Sundberg C, Juthberg R, Olesen A, Guo L, Persson NK, Ackermann PW. Transcutaneous Electrical Nerve Stimulation Integrated into Pants for the Relief of Postoperative Pain in Hip Surgery Patients: A Randomized Trial. Pain Res Manag. 2024 Jun 27;2024:6866549. doi: 10.1155/2024/6866549. eCollection 2024. PMID 39145150